CLINICAL TRIAL: NCT04770246
Title: A Phase 2 Study of TAS-117 in Patients With Advanced Solid Tumors Harboring Germline PTEN Inactivating Mutations
Brief Title: TAS-117 in Patients With Advanced Solid Tumors Harboring Germline PTEN Mutations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor had decided to terminate this clinical trial due to an insufficient rate of accrual of patients.
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS-117-201; 2020-004770-22 (EudraCT Number)
Record Dates: First submitted 2021-02-16; First posted 2021-02-25 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Advanced or Metastatic Solid Tumors Irrespective of Gene Alterations; Advanced or Metastatic Solid Tumors With Germline PTEN Inactivating Mutations
Keywords: TAS-117; AKT inhibitor; Allosteric inhibitor; Advanced solid tumor; Metastatic solid tumor; PTEN; Germline PTEN; Inactivating mutation; Adolescent patients; Adult patients
MeSH Terms: conditions — Neoplasm Metastasis | interventions — 3-amino-1-methyl-3-(4-(3-phenyl-5H- imidazo(1,2-c)pyrido(3,4-e)(1,3)oxazin-2-yl)phenyl)cyclobutanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TAS-117 Dose Escalation Daily Dose Regimen (Part A: safety lead-in) (Experimental): Advanced or metastatic solid tumors irrespective of gene alterations
  Interventions: Drug: TAS-117
- TAS-117 Dose Escalation Intermittent Dose Regimen (Part A: safety lead-in) (Experimental): Advanced or metastatic solid tumors irrespective of gene alterations
  Interventions: Drug: TAS-117
- TAS-117 Dose and Regimen Confirmation (Part A: safety lead-in) (Experimental): Advanced or metastatic solid tumors with germline PTEN inactivating mutations
  Interventions: Drug: TAS-117
- TAS-117 Phase 2 (Part B) (Experimental): Advanced or metastatic solid tumors with germline PTEN inactivating mutations
  Interventions: Drug: TAS-117

INTERVENTIONS:
Drug: TAS-117 — TAS-117 will be dosed orally every day on a 21-day cycle
  Arms: TAS-117 Dose Escalation Daily Dose Regimen (Part A: safety lead-in)
Drug: TAS-117 — TAS-117 will be dosed intermittently on a 21-day cycle
  Arms: TAS-117 Dose Escalation Intermittent Dose Regimen (Part A: safety lead-in)
Drug: TAS-117 — TAS-117 will be dosed orally every day or intermittently on a 21-day cycle
  Arms: TAS-117 Dose and Regimen Confirmation (Part A: safety lead-in)
Drug: TAS-117 — TAS-117 will be dosed orally every day or intermittently on a 21-day cycle
  Arms: TAS-117 Phase 2 (Part B)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and antitumor activity of TAS-117 in patients with advanced or metastatic solid tumors (excluding primary brain tumors) harboring germline PTEN inactivating mutations.

DETAILED DESCRIPTION:
Study TAS-117-201 is an open-label, single-arm Phase 2 study evaluating the efficacy, safety, tolerability, pharmacokinetics, and pharmacodynamics of TAS-117 in patients with advanced or metastatic solid tumors harboring germline PTEN inactivating mutations. The study will be conducted in two parts:

* Part A: Safety lead-in (Dose Escalation and Dose Regimen Confirmation)
* Part B: Single-arm Phase 2 study

Patients will receive TAS-117 orally every day or intermittently on a 21-day cycle

* Part A (Dose Escalation): up to 36 adult patients with advanced or metastatic solid tumors (excluding primary brain tumors) irrespective of gene alterations. The Dose Escalation consists of 2 cohorts: Daily Dose Regimen and Intermittent Dose Regimen.
* Part A (Dose Regimen Confirmation): approximately 6 adult or adolescent patients with advanced or metastatic solid tumors (excluding primary brain tumors) harboring germline PTEN inactivating mutations
* Part B (Phase 2): approximately 54 adult or adolescent patients with advanced or metastatic solid tumors (excluding primary brain tumors) harboring germline PTEN inactivating mutations

Treatment will continue until disease progression, unacceptable toxicity, or any other of the criteria for treatment discontinuation is met. For patients who discontinue treatment for reasons other than disease progression, tumor assessments should be continued until radiologic disease progression is documented or until initiation of subsequent new anticancer therapy (whichever occurs first).

Patients will be followed for survival every 12 weeks (±2 weeks) until survival events (deaths) have been reported for 75% of enrolled patients or the study is terminated early by the Sponsor.

ELIGIBILITY:
Inclusion Criteria

1. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
2. Dose Escalation in Part A

   1. ≥18 years of age.
   2. Histologically or cytologically confirmed advanced or metastatic solid tumors
   3. Has progressed after standard treatment for advanced or metastatic disease or was intolerant to or ineligible for available standard therapies.
   4. Patients with solid tumors irrespective of gene alterations.
   5. Patients with at least one measurable or non-measurable lesion per RECIST1.1
3. Dose and Regimen Confirmation in Part A and Phase 2 (Part B)

   1. ≥12 years of age. Patients age ≥12 and <18 years must have a body weight of ≥40 kg.
   2. Histologically confirmed advanced or metastatic solid tumors.
   3. Has progressed after standard treatment for advanced or metastatic disease or was intolerant or ineligible to available standard therapies.
   4. Patients with locally confirmed germline PTEN inactivating mutations determined from a blood sample.
   5. Patients with at least one measurable lesion per RECIST 1.1.

Exclusion Criteria

1. History or current evidence of interstitial lung disease that requires steroid medication.
2. Current evidence of diabetes mellitus that requires insulin therapy.
3. Prior treatment with PI3K/AKT/mTOR pathway inhibitors.
4. Patients with primary brain tumor.
5. Patients with meningeal carcinomatosis, leptomeningeal carcinomatosis, spinal cord compression, or symptomatic or unstable brain metastasis.
6. Currently receiving chronic corticosteroid therapy of ≥10 mg/day of prednisone or its equivalent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events and dose-limiting toxicities (safety and tolerability) and MTD of TAS-117 in Part A | 21 days for DLT evaluation, approximately 7 months for the others
  Number of patients with abnormal laboratory values, treatment emergent AEs, abnormal vital signs and ECG, and Dose-limiting toxicities (DLTs)
Recommended Phase 2 Dose (RP2D) of TAS-117 in Part A | 21 days for DLT evaluation, approximately 7 months for the others
Objective Response Rate (ORR) in Part B (including all patients with germline PTEN mutations in Part A) | Approximately 6 months
  ORR, defined as the proportion of patients experiencing a best overall response of CR or PR per RECIST 1.1.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety) in Part B | Approximately 7 months
  Number of patients with abnormal laboratory values, treatment-emergent AEs, abnormal vital signs and ECG
Disease Control Rate (DCR) | Approximately 6 months
  DCR, defined as the proportion of patients experiencing a best overall response of stable response (SD), PR, or complete response (CR).
Duration of Response (DOR) | Approximately 6 months
  DOR, defined as the time from the first documentation of response (CR or PR) to the first documentation of objective tumor progression or death due to any cause, whichever occurs first.
Progression Free Survival (PFS) | Approximately 6 months
  PFS, defined as the time from date of the first dose of study treatment to the date of disease progression based on Investigator assessment of radiographic images or death, whichever occurs first.
Overall Survival (OS) | Approximately 12 months
  OS, defined as the time from the date of first dose to the death date.
Pharmacokinetics (PK) profile of TAS-117 in Part A | 21 days
  maximum plasma concentration (Cmax)
Pharmacokinetics (PK) profile of TAS-117 in Part A | 21 days
  area under the plasma concentration-time curve (AUC)
Pharmacokinetics (PK) profile of TAS-117 in Part A | 21 days
  time to reach maximum plasma concentration (Tmax)
Pharmacokinetics (PK) profile of TAS-117 in Part A | 21 days
  terminal elimination half-life (T1/2)
Pharmacodynamics (PD) profile of TAS-117 in Part A | 21 days
  Evaluate Total and Phosphorylated AKT and PRAS40

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Lerner Research Institute, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Medical University of Vienna, Vienna, Austria
- Institut Gustave Roussy, Villejuif, Île-de-France Region, France
- Sarah Cannon Research Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodon J, Funchain P, Laetsch TW, Arkenau HT, Hervieu A, Singer CF, Murciano-Goroff YR, Chawla SP, Anthony K, Yamamiya I, Liu M, Halim AB, Benhadji KA, Takahashi O, Delaloge S. A phase II study of TAS-117 in patients with advanced solid tumors harboring germline PTEN-inactivating mutations. Future Oncol. 2022 Sep;18(30):3377-3387. doi: 10.2217/fon-2022-0305. Epub 2022 Aug 30. PMID 36039910